CLINICAL TRIAL: NCT01642056
Title: Therapeutic Trial of EPI -743 In Patients With Disorders of Energy Utilization or Oxidation-Reduction
Brief Title: EPI-743 for Metabolism or Mitochondrial Disorders
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 120161; 12-HG-0161
Record Dates: First submitted 2012-07-14; First posted 2012-07-17 (Estimated); Results first posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2019-12-09

CONDITIONS: Mitochondrial Disease; Neurology; Myopathy
Keywords: Oxidative Stress; Oxidative Phosphorylation; Mitochondrial Disease
MeSH Terms: conditions — Mitochondrial Diseases; Muscular Diseases | interventions — alpha-tocotrienol quinone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EPI-743, then Placebo (Experimental): Received EPI-743, 15mg/kg up to a maximum dose of 200 mg orally or via gastric tube three times daily with meals, then placebo three times daily orally or via gastric tube with meals. EPI-743 is structurally related to Vitamin E and can be broadly classified as an antioxidant.
  Interventions: Drug: EPI-743; Drug: Placebo
- Placebo, then EPI-743 (Placebo Comparator): Received Placebo three times daily orally or via gastric tube with meals, then EPI-743, 15mg/kg up to a maximum dose of 200 mg three times daily orally or via gastric tube with meals. EPI-743 is structurally related to Vitamin E and can be broadly classified as an antioxidant.
  Interventions: Drug: EPI-743; Drug: Placebo

INTERVENTIONS:
Drug: EPI-743 — This medication is used to treat disorders of energy metabolism such as mitochondrial diseases. It does not correct the inherited disorder of energy metabolism or mitochondrial diseases. EPI-743 is structurally related to Vitamin E and can be broadly classified as an antioxidant.
Drug: Placebo

SUMMARY:
Background:

* Mitochondria are the parts of cells that help produce energy. Metabolism is the process by which the body uses energy to help cells grow and reproduce. Metabolic and mitochondrial disorders affect the body s ability to produce and store energy. These disorders can cause a wide variety of problems, but most often they affect the muscles and the brain, where energy requirements are high. Treatment is difficult because the exact source of the problem is hard to detect.
* EPI-743 is a new drug that is based on vitamin E. Tests have shown that it can help improve the function of cells with mitochondrial problems. It may be able to treat people with genetic disorders that affect metabolism and mitochondria.

Objectives:

- To see if EPI-743 can improve energy production and use in people with mitochondrial or metabolic disorders.

Eligibility:

- Children between 2 and 11 years of age who have metabolic or mitochondrial problems.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected.
* The study will last about 13 months. Participants will have seven 3- to 5-day inpatient study visits about 3 months apart.
* Participants will take either EPI-743 or a placebo for the first 6 months of the study. After 6 months, there will be a 1-month rest period. Then, those who received EPI-743 in the first 6 months will take the placebo for the next 6 months. Those who had the placebo will take EPI-743.
* During each inpatient study visit, participants will have a physical exam. A 24-hour urine collection will be obtained. Blood samples will also be taken. Imaging studies and other tests may be performed as directed by the study researchers.

DETAILED DESCRIPTION:
The clinical manifestations of disorders of energy metabolism and defects in oxidation/reduction are similar because the basic defect involves the inability to transfer electrons. The same is true for many mitochondrial diseases. Affected patients exhibit a wide variety of signs and symptoms, but the most frequent and earliest dysfunctions occur in the muscle and brain, where energy requirements are high. The diagnosis of this type of defect is problematic because of the nonspecific and protean clinical manifestations of these disorders. Treatment is equally challenging, since the exact locus of the primary defect generally remains enigmatic. As a consequence, physicians rely upon generic cocktails of vitamin co-factors or endogenous intermediates intended to enhance mitochondrial electron transport, diminish the damage of reactive oxygen species, and promote energy production. The field is such a morass that, in general, it calls for trial-and-error treatment based upon empiric data. Edison Pharmaceuticals, Inc, has developed an in vitro assay that utilizes patient fibroblasts to model the innate susceptibility to oxidative stress caused by the disorders of energy metabolism and oxidation/reduction. The assay system also determines if the cells respond with increased viability to an IND drug called EPI-743. We propose a clinical trial that enrolls 20 children who meet three criteria. First, they must have a disorder that, based upon studies performed in a clinical protocol such as 76-HG-0238 ("Diagnosis and Treatment of Patients with Inborn Errors of Metabolism and Other Genetic Disorders"), is consistent with a defect in energy metabolism or oxidation/reduction. Second, their cultured fibroblasts must exhibit a defect in the ability to withstand oxidant stress. Third, their fibroblasts must respond to EPI-743 in vitro by showing improved viability under conditions of oxidative stress. This protocol is a double-blind, placebo-controlled crossover study with 6-month periods of treatment and a two-month washout period. Patients will be admitted to the NIH Clinical Center for 2-5 days every 3 months. The primary outcome measure will be quality of life based upon the Newcastle Paediatric Mitochondrial Disease Scale (NPMDS) for ages 2-11 years; parts IIII

will be evaluated separately from part IV. Secondary outcome measures will be tailored to each patient's laboratory, imaging, and clinical abnormalities. Results while receiving EPI-743 will be compared to results while receiving placebo; both repeated measures analyses and Student's t test will be employed.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion criteria involve enrollment in protocol 76-HG-0238, Diagnosis and Treatment of Patients with Inborn Errors of Metabolism and Other Genetic Disorders . In addition, patients must:

* Be 2-11 years of age
* Manifest clinical findings of a neuromuscular disease with a component of impaired energy or oxidation/reduction. Typical symptoms would include hypotonia, dystonia, or seizures.
* Have a disorder that is untreatable or poorly treatable.
* Have cultured fibroblasts that exhibit reduced viability under conditions of oxidative stress, compared to age matched control fibroblasts.
* Have cultured fibroblasts that achieve at least 80% viability rescue with EPI-743 at 1micromolar upon exposure to oxidative stress and that have a half maximal effective concentration of EPI-743 of less than or equal to 50 nanomolar.
* Be willing to abstain from initiating the use of dietary supplements and nonprescribed medications, foods or beverages or bars fortified with coenzyme Q(10), vitamin E, super fortified functional foods or beverages, and idebenone.
* Be able to travel to the Clinical Center for at least 8 visits.

EXCLUSION CRITERIA:

* Age < 2 years or >11 years
* Diagnosis of mitochondrial diseases benefiting from treatment and at risk from being moved to placebo
* Allergy to EPI-743 or sesame oil
* Hepatic insufficiency with liver function tests greater than 3-times the upper limit of normal
* Renal insufficiency requiring dialysis
* Significant malabsorption of fats precluding drug absorption
* Allergy to vitamin E
* Significant coagulation abnormalities as evidenced by abnormal PT/PTT tests
* Severe end-organ hypo-perfusion syndrome secondary to cardiac failure resulting in lactic acidosis
* Ventilator-dependence
* Chronic pancreatitis
* Clinical history of bleeding requiring ongoing medical management
* Abnormal red cell parameters requiring ongoing medical management besides iron supplementation
* A platelet disorder
* Neutrophils less than 500 mm3

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2012-09-01; Primary Completion 2019-09-24 (Actual); Study Completion 2019-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William A Gahl, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Shrader WD, Amagata A, Barnes A, Enns GM, Hinman A, Jankowski O, Kheifets V, Komatsuzaki R, Lee E, Mollard P, Murase K, Sadun AA, Thoolen M, Wesson K, Miller G. alpha-Tocotrienol quinone modulates oxidative stress response and the biochemistry of aging. Bioorg Med Chem Lett. 2011 Jun 15;21(12):3693-8. doi: 10.1016/j.bmcl.2011.04.085. Epub 2011 Apr 24. PMID 21600768
- [Background] Sadun AA, Chicani CF, Ross-Cisneros FN, Barboni P, Thoolen M, Shrader WD, Kubis K, Carelli V, Miller G. Effect of EPI-743 on the clinical course of the mitochondrial disease Leber hereditary optic neuropathy. Arch Neurol. 2012 Mar;69(3):331-8. doi: 10.1001/archneurol.2011.2972. PMID 22410442
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-HG-0161.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 20 subjects were consented. One subject died during first intervention due to progression of disease. Three subjects did not complete the second intervention.
Period: First Intervention
Arm/Group | EPI-743, Then Placebo | Placebo, Then EPI-743
Started | 10 | 10
Completed | 9 | 10
Not Completed | 1 | 0
Period: Second Intervention
Arm/Group | EPI-743, Then Placebo | Placebo, Then EPI-743
Started | 9 | 10
Completed | 8 | 8
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EPI-743, Then Placebo | Placebo, Then EPI-743 | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 10 | 20
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 7 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 9 | 9 | 18
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 4 | 9 | 13
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Newcastle Paediatric Mitochondrial Disease Scale (NPMDS) Part I-III, Baseline
Description: NPMDS is a semi-quantitative clinical rating scale that evaluates the progression of mitochondrial disease in pediatric patients.
  The NPMDS scale provides an assessment of the progression of mitochondrial disease. Scores from Parts I-III are added to get a value between 0 and 130, with higher scores representing more severe disease.
Time Frame: Baseline - Day 0
Population: Participants who who had treatment intervention in phase I. The outcome measures were analyzed separately by arm and phase, not by combining results by intervention across phases, due to the progressive nature of the underlying disease.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | EPI-743, Then Placebo | Placebo, Then EPI-743
Number analyzed (Participants) | 10 | 10
Units on a scale | 23.9 (2.8) | 20.4 (3.7)

2. Primary Outcome: Newcastle Paediatric Mitochondrial Disease Scale (NPMDS) Part I-III, 6 Months
Description: as for outcome 1
Time Frame: 6 months
Population: (Participants who who had treatment intervention in phase I. The outcome measures were analyzed separately by arm and phase, not by combining results by intervention across phases, due to the progressive nature of the underlying disease.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | EPI-743, Then Placebo | Placebo, Then EPI-743
Number analyzed (Participants) | 9 | 10
Units on a scale | 27.1 (2.7) | 20.2 (3.8)

3. Primary Outcome: Newcastle Paediatric Mitochondrial Disease Scale (NPMDS) Part I-III, Post Washout
Description: as for outcome 1
Time Frame: 8 month - Post washout
Population: Participants who received treatment in phase II. The outcome measures were analyzed separately by arm and phase, not by combining results by intervention across phases, due to the progressive nature of the underlying disease.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | EPI-743, Then Placebo | Placebo, Then EPI-743
Number analyzed (Participants) | 9 | 10
Units on a scale | 27.1 (3.5) | 18.3 (3.6)

4. Primary Outcome: Newcastle Paediatric Mitochondrial Disease Scale (NPMDS) Part I-III, 14 Months
Description: as for outcome 1
Time Frame: 14 months
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | EPI-743, Then Placebo | Placebo, Then EPI-743
Number analyzed (Participants) | 8 | 8
Units on a scale | 26 (3.3) | 15.8 (3.7)

ADVERSE EVENTS:
Time Frame: 14 Months
Groups:
- EPI-743: Received EPI-743, 15mg/kg up to a maximum dose of 200 mg orally or via gastric tube three times daily with meals. EPI-743 is structurally related to Vitamin E and can be broadly classified as an antioxidant.
- Placebo: Received Placebo three times daily orally or via gastric tube with meals.
Arm/Group | EPI-743 | Placebo
All-Cause Mortality (participants affected / at risk) | 1/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 3/20 | 4/19
Other Adverse Events (participants affected / at risk) | 17/20 | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EPI-743 (N=20) | Placebo (N=19)
Hyperthermia (General disorders) | 0 | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (3) | 0
Status epilepticus (Nervous system disorders) | 1 (1) | 0
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Hospitalisation (Surgical and medical procedures) | 2 (3) | 4 (6)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EPI-743 (N=20) | Placebo (N=19)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 (3)
Polycythaemia (Blood and lymphatic system disorders) | 2 (3) | 5 (5)
Tinnitus (Ear and labyrinth disorders) | 0 | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0
Goitre (Endocrine disorders) | 1 (1) | 0
Hypercalcaemia (Endocrine disorders) | 0 | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 2 (2)
Hypothyroidism (Endocrine disorders) | 3 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 | 2 (2)
Gastroenteritis viral (Gastrointestinal disorders) | 1 (1) | 0
Nausea (Gastrointestinal disorders) | 0 | 1 (1)
Pharyngitis (Gastrointestinal disorders) | 0 | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 4 (5)
Fatigue (General disorders) | 0 | 2 (2)
Hyperthermia (General disorders) | 0 | 6 (6)
Influenza like illness (General disorders) | 0 | 1 (1)
Hyperammonaemia (Hepatobiliary disorders) | 1 (1) | 0
Activated partial thromboplastin time prolonged (Investigations) | 3 (4) | 5 (6)
Alanine aminotransferase increased (Investigations) | 4 (7) | 4 (5)
Amylase increased (Investigations) | 1 (1) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 4 (5) | 4 (6)
Blood albumin decreased (Investigations) | 0 | 2 (3)
Blood alkaline phosphatase increased (Investigations) | 2 (3) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 10 (14) | 6 (10)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 1 (2)
International normalised ratio increased (Investigations) | 1 (1) | 0
Lipase increased (Investigations) | 1 (1) | 0
Lymphocyte count increased (Investigations) | 0 | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 2 (2)
Platelet count decreased (Investigations) | 1 (1) | 2 (2)
Prothrombin time prolonged (Investigations) | 1 (1) | 0
Red blood cell sedimentation rate increased (Investigations) | 1 (1) | 0
White blood cell count decreased (Investigations) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 | 1 (1)
Hyperbilirubinaemia (Metabolism and nutrition disorders) | 1 (1) | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 2 (2) | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 (1)
Psychomotor hyperactivity (Psychiatric disorders) | 0 | 1 (1)
Violence-related symptom (Psychiatric disorders) | 0 | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Upper respiratory tract irritation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0

LIMITATIONS AND CAVEATS:
All 20 randomized patients were included in the model to assess baseline characteristics. Of the 20 randomized, 19 provided 6-month outcomes (10 placebo, 9 treatment), who then crossed over their treatments and provided 8-month baseline scores. Of these, 16 provided 14-month outcomes (8 who had crossed over to treatment, and 8 who had crossed over to placebo).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT01642056/Prot_SAP_000.pdf